CLINICAL TRIAL: NCT04018755
Title: Open-label Pilot Study of the Effects of Anakinra in Mucopolysaccharidosis (MPS) III
Brief Title: Open-label Study of Anakinra in MPS III
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lynda E Polgreen (Other)
Collaborators: Cure Sanfilippo Foundation (Unknown); Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor-Investigator, Lynda E Polgreen, Investigator/Associate Professor, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Organization: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31834-01
Record Dates: First submitted 2019-07-01; First posted 2019-07-12 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Mucopolysaccharidosis III
MeSH Terms: conditions — Mucopolysaccharidosis III | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment (Experimental): anakinra 100 mg subcutaneous once daily
  Interventions: Biological: anakinra

INTERVENTIONS:
Biological: anakinra — anakinra single-use prefilled glass syringes
  Other Names: Kineret

SUMMARY:
Sanfilippo syndrome, or mucopolysaccharidosis type III (MPS III), is a disorder of metabolism, associated with insufficient production of a lysosomal enzyme needed for normal cell function. As a consequence of the cellular dysfunction, patients with this disorder develop progressive, irreversible neurodegeneration. Sadly, to date no evidence-based treatments are available.

Inflammation has been connected with disease pathogenesis in the MPS disorders. Therapies aimed at decreasing inflammation are currently being studied in many MPS disorders and benefits in both brain and other parts of the body have been reported.Decreasing interleukin-1 (IL-1) in an animal model of MPS III showed benefits in brain disease and behavior. Thus, we think that anakinra (Kineret), which decreases IL-1 levels in the body, will improve behavioral and other problems in children with MPS III.

Anakinra is approved by the FDA for treatment of rheumatoid arthritis (RA) and neonatal-onset multisystem inflammatory disease (NOMID). It is not approved for any MPS disorder.

The design of this study is an open-label, single center, pilot study of 20 participants with MPS III. There will be an initial screening visit, followed by an 8-week observational period, then a 36-week treatment period, and finally another 8-week observational period to determine any effects of withdrawal from the treatment.

During visits the participants will undergo a medical history, a physical examination, and anthropometric measurements. Blood, urine, and stool will be collected for biomarker levels and safety laboratory studies. Questionnaires will be completed with questions related to behavior, stooling, sleep, and activities of daily living. Seizure and movement disorders will be monitored as well.

The most common risks of receiving anakinra, based on RA and NOMID experience, include local injection site reactions, headache, nausea, vomiting, arthralgia, and flu-like symptoms. The most serious potential risk is a serious infection and neutropenia. However, because so few people with MPS have been treated with anakinra, all the risks related to MPS patients receiving anakinra are not currently known. Additional risks related to taking part in the study include some pain, bruising, and/or bleeding due to blood draws/peripheral IV placement, and discomfort with completing some of the questionnaires.

The expected potential direct benefits include, but are not limited to, improved behavior, sleep, stooling, communication, mood, and gait; as well as decreased seizure frequency, disordered movement and fatigue. However, there is no guarantee that participants will get any benefit from being in this study.

ELIGIBILITY:
Inclusion Criteria:

* MPS III
* ≥ 4 years of age
* Patient or parent/legal guardian is able and willing to provide informed consent. For patients 7 to 17 years of age, assent must also be provided when cognitively possible.
* If on Genistein, must have been on a stable dose for 6 months prior to enrollment
* If on melatonin or other sleep medications, must have been on stable doses for the past 3 months

Exclusion Criteria:

* Currently enrolled in another ongoing clinical treatment trial
* Previous or current treatment with anakinra, canakinumab or any other IL-1 inhibitor.
* Use of the following therapies prior to enrollment:

  * Narcotic analgesics within 24 hours prior to enrollment.
  * Tocilizumab, dapsone or mycophenolate mofetil within 3 weeks prior to enrollment.
  * Etanercept, leflunomide, thalidomide, or cyclosporine or intraarticular, intramuscular, intravenous, or oral administration of glucocorticoids within 4 weeks prior to enrollment.
  * Intravenous immunoglobulin (IVIG), adalimumab, or methotrexate within 8 weeks prior to enrollment.
  * Infliximab, 6-mercaptopurine, azathioprine, cyclophosphamide or chlorambucil within 12 weeks prior to enrollment.
  * Rituximab within 26 weeks prior to enrollment
* Live vaccines within 1 month prior to enrollment.
* Known presence or suspicion of active, chronic or recurrent serious bacterial, fungal or viral infections, including tuberculosis, HIV infection or hepatitis B or C infection.
* Clinical evidence of liver disease or liver injury as indicated by presence of abnormal liver tests:

  * AST or ALT > 5 x ULN, or
  * AST or ALT > 3 x ULN accompanied by elevated bilirubin >2 x ULN.
* Presence of severe renal function impairment (estimated creatinine clearance < 30 mL/min/1.73m2).
* Presence of neutropenia.
* History of malignancy.
* Known hypersensitivity to E coli-derived proteins, or any components of Kineret® (anakinra).
* Pregnant or lactating women.
* Current active infection;
* History of serious opportunistic infection (e.g., bacterial [Legionella and Listeria]; tuberculosis [TB]; invasive fungal infections; or viral, parasitic, and other opportunistic infections);
* Positive TB skin test, positive Quantiferon-TB Gold TB test, positive chest X-ray, or a recent exposure to TB
* Requirement for live vaccine exposure that would be expected to occur during the time frame of the study

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2022-07-17 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
The percent of participants who required an increase in anakinra dose from 100 mg SC daily to 200 mg SC daily at Week 8 or Week 16 | up to 8 weeks of treatment
  Need for dose escalation was determined by within individual change over an 8-week treatment period compared to change over the 8-week pre-treatment observational period in the 2 most bothersome symptoms for each enrolled patient chosen by their caregiver and selected from 6 suverys included in the Multi-domian Responder Index (MDRI). These surveys were:
  * Sanfilippo Behavior Rating Scale (SBRS)
  * Child Sleep Health Questionnaire (CSHQ)
  * Autism Parenting Stress Index (APSI)
  * PROMIS Fatigue - Parent Proxy Custom Short Form
  * Movement disorder - parent reported frequency, duration, and severity (7-day log)
  * Non-communicating Children's Pain Checklist-Revised (NCCPC-R)

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Polgreen, MD, MS, Principal Investigator — The Lundquist Institute at Harbor-UCLA Medical Center
Locations (1):
- The Lundquist Institute at Harbor-UCLA Medical Center, Torrance, California, United States

REFERENCES:
- [Derived] Polgreen LE, Chen AH, Pak Y, Luzzi A, Morales Garval A, Acevedo J, Bitan G, Iacovino M, O'Neill C, Eisengart JB. Anakinra in Sanfilippo syndrome: a phase 1/2 trial. Nat Med. 2024 Sep;30(9):2473-2479. doi: 10.1038/s41591-024-03079-3. Epub 2024 Jun 21. PMID 38907160